CLINICAL TRIAL: NCT07221734
Title: Randomised, Multicentre, Multinational, Double-Blind Integrated Study to Compare the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of MB11 (Proposed Nivolumab Biosimilar) Versus EU-/US-Opdivo® in Subjects With Previously Untreated Advanced (Unresectable or Metastatic) Melanoma (LEON Study)
Brief Title: Study to Compare Pharmacokinetics, Efficacy, Safety, and Immunogenicity of MB11 Versus EU-/US-Opdivo® in Subjects With Previously Untreated Advanced [Unresectable or Metastatic] Melanoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB11-C-01-25
Record Dates: First submitted 2025-10-06; First posted 2025-10-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced (Unresectable or Metastatic) Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB11 (Proposed Nivolumab Biosimilar) (Experimental)
  Interventions: Drug: MB11 (Proposed Nivolumab Biosimilar)
- EU-Opdivo® (Active Comparator)
  Interventions: Drug: EU-Opdivo®
- US- sourced Opdivo® (Active Comparator)
  Interventions: Drug: US- sourced Opdivo®

INTERVENTIONS:
Drug: MB11 (Proposed Nivolumab Biosimilar) — During fist 12 cycles: 3 mg/kg IV infusion, over 30 minutes, Q2W. On Cycle 13 onwards: 3 mg/kg IV infusion, over 30 minutes, Q2W or 240 mg flat dose Q2W dosing
  Arms: MB11 (Proposed Nivolumab Biosimilar)
Drug: EU-Opdivo® — During fist 12 cycles: 3 mg/kg IV infusion, over 30 minutes, Q2W. On Cycle 13 onwards: 3 mg/kg IV infusion, over 30 minutes, Q2W or 240 mg flat dose Q2W dosing
  Arms: EU-Opdivo®
Drug: US- sourced Opdivo® — During fist 12 cycles: 3 mg/kg IV infusion, over 30 minutes, Q2W. On Cycle 13 onwards: 3 mg/kg IV infusion, over 30 minutes, Q2W or 240 mg flat dose Q2W dosing
  Arms: US- sourced Opdivo®

SUMMARY:
This is a randomised, multicentre, multinational, double-blind, integrated study to sompare the pharmacokinetics, efficacy, safety, and immunogenicity of MB11 versus Opdivo® in subjects with previously untreated advanced (unresectable or Metastatic) Melanoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent (or adulthood where the legalage of majority in the country is established >18 years).
2. Body weight ≥50 kg at baseline.
3. Signed informed consent must be obtained before initiation of any study-specific procedures or treatment.
4. ECOG performance status of 0 or 1.
5. Life expectancy for at least 3 months.
6. Untreated, histologically confirmed advanced unresectable Stage III or Stage IV melanoma, as per AJCC 8th Edition staging system. Prior melanoma systemic therapy for earlier stages is allowed for patients who have been disease-free for at least 1 year after end of therapy, except if therapy included use of prohibited medications. Prior use of immune therapies (adjuvant or neoadjuvant) is not allowed as per Exclusion Criteria #2.
7. At least 1 measurable disease lesion by CT or MRI per RECIST v1.1 criteria.
8. Tumour tissue from an unresectable or metastatic site of disease, collected within 90 days prior to randomisation, must be available and provided for PD-L1 testing. All samples must be classified as PD-L1 positive (≥1% to <5% or ≥5%). If only the old sample >90 days is available and there is no possibility of having a new biopsy sample, then the subject will be excluded.
9. In the case of prior palliative radiotherapy (on metastatic lesions), this must have been completed at least 2 weeks prior to the study drug administration. No adjuvant radiation therapies are allowed.
10. Any BRAF mutation status is allowed (BRAF-mutated, BRAF wild-type or non-mutated, or BRAF status unknown).
11. Adequate organ function (bone marrow, hepatic, renal, haematologic, endocrine, and coagulation function) should be demonstrated during the screening period. This is defined as:

    1. Haematologic function: absolute neutrophil count ≥1.5 × 109/L, platelets 9≥100 × 10 /L, and haemoglobin ≥9 g/dL.

       ** Subjects should not have received RBC transfusion prior to 14 days beforescreening labs.
    2. Renal function: serum creatinine level ≤1.5 × ULN or calculated CrCl ≥60 mL/min (using the Cockcroft-Gault formula).
    3. Liver function: total bilirubin level ≤1.5 × ULN (except subjects with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL), albumin level ≥LLN, AST/ALT ≤2.5 × ULN (≤5 × ULN for subjects with liver metastases).
    4. Endocrine function: TSH within normal limits. If TSH is not within normal limits, the subject may still be eligible if T3 and free T4 are within normal limits.
    5. Coagulation: INR and aPTT ≤1.5 × ULN unless the subject is receiving anticoagulant therapy. Subjects on anticoagulant therapy must be on a stable anticoagulation regimen and have an INR not above the target therapeutic range for the 14 days preceding the start of the study drug.
12. Female subjects of childbearing potential and their partners, as well as male subjects with female partners of childbearing potential and their partners, must agree to adhere to the use of a highly effective method of contraception during the study and for at least 5 months after the last dose of nivolumab. Refer to Appendix 15.1 for contraception guidance.
13. Non-fertile females can be included.

Exclusion Criteria:

1. Subjects receiving any prior systemic therapy for advanced, unresectable, or metastatic Stage III or Stage IV melanoma (except for palliative radiotherapy, in accordance with Inclusion Criteria #9).
2. Subjects receiving any prior immunotherapy (regardless of the melanoma stage), such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-LAG or anti-CTLA-4 therapy (including ipilimumab or any other antibody or drug that specifically targets costimulation of T-cells or immune checkpoints) and/or BRAF-targeted therapy.
3. Participation in another clinical study or treatment with another investigational agent within 4 weeks or 5 elimination half-lives prior to randomisation (whichever is longer)
4. Brain metastases or leptomeningeal metastases. A negative brain imaging of less than 90 days prior to screening is required.
5. Peritoneal melanomatosis.
6. Ocular melanoma, mucosal melanoma and acral lentiginous melanoma.
7. History of another malignancy or a concurrent malignancy. Exceptions include subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
8. Active autoimmune disease that has required systemic treatment in the last 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin or physiological corticosteroid replacement therapy for pituitary or adrenal insufficiency [daily prednisone at a dose of ≤10 mg or equivalent]) is not considered a form of systemic treatment.
9. Subjects with hyperthyroidism or hypothyroidism are excluded but those subjects who are stable on hormone replacement will be allowed.
10. Any diagnosis of immunodeficiency, systemic steroid therapy (replacement therapy outlined in Exclusion Criteria #8, inhaled, intranasal, intraocular, or topical steroids are allowed) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug.
11. Any major surgery (eg, hip or spine surgery) less than 28 days prior to the first dose of the study drug.
12. Having received a solid organ/tissue allogeneic or haematopoietic transplant.
13. History and/or current interstitial lung disease or pneumonitis (non-infectious) requiring oral or IV steroids or another immunosuppressive drug.
14. Any active or previous infection requiring therapy (oral or systemic) within 30 days prior to the first dose of the study drug.
15. Have received or are about to receive a live virus vaccination within 30 days prior to the first dose of the study drug. Seasonal flu and COVID-19 vaccines that do not contain live virus are permitted.
16. Known active TB or untreated latent TB.
17. Positive serology for human immunodeficiency virus (HIV 1/2), hepatitis B (HBsAg positive and/or HBcAb positive, and HBV DNA positive, refer to Section 8.3.2.1) or hepatitis C (HCVAb positive and HCV RNA positive). In addition, subjects with untreated positive serology for Strongyloides spp will be excluded.
18. At the time of signing the informed consent, the subject is a regular user (including "recreational use") of any illicit drug or have a recent history (within the past year) of substance abuse (including alcohol).
19. Be pregnant or lactating or expecting to conceive during the study or up to 5 months after the last dose of the study drug.
20. Immediate family member who is at the research site or sponsoring staff who is directlyninvolved in this study.
21. Inability to comply with protocol procedures and/or any other acute or chronic medical condition that may increase the risk for the subject associated with study participation or study drug administration, that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the Pharmacokinetic (PK) bioequivalence between MB11 and EU/ US-Opdivo. | Week 1 - Week 24
  Area under the concentration-time curve (AUC) between Cycle 1 and Cycle 2 (AUC from time 0 to 504 hours postdose [AUC0-336]. AUC at steady state (AUCss) between Cycle 8 and Cycle 9.
To demonstrate the efficacy equivalence of MB11 and Opdivo® administered as first-line treatment in adult subjects with untreated, unresectable, or metastatic Stage III or Stage IV melanoma | Week 1 - Week 24
  Best Overall Response (BOR), prior to permanent treatment discontinuation, prior to use of other anti-cancer therapies and by 24 weeks after Day 1

SECONDARY OUTCOMES:
To compare the efficacy of MB11 with Opdivo based on other efficacy parameters and timepoints over the study period. | Week 1 - Week 52
  Progression-free survival (PFS)
To compare the efficacy of MB11 with Opdivo based on other efficacy parameters and timepoints over the study period. | Week 1 - Week 52
  Duration of response (DOR)
To compare the efficacy of MB11 with Opdivo based on other efficacy parameters and timepoints over the study period. | Week 1 - Week 52
  Overall survival (OS)
.To compare the PK profile based on other PK parameters and timepoints (not covered by the primary PK endpoints) of MB11 as compared with Opdivo® over the study period. | Week 1 - Week 52
  Maximum concentration (Cmax), Minimum concentration (Ctrough),
To assess the safety and tolerability of MB11 as compared with Opdivo® | Week 1 - Week 52
  Treatment-emergent adverse events (TEAEs)
To assess the immunogenicity of MB11 as compared with Opdivo® | Week 1 - Week 52
  Anti-drug antibodies (ADAs) and Neutralizing antibodies (NAbs) in ADA-positive samples

CONTACTS AND LOCATIONS:
Locations (19):
- Site 111003, Funchal, Portugal
- Ukraine (18):
  - Site 117015, Chernivtsi
  - Site 117005, Ivano-Frankivsk
  - Site 117002, Kyiv
  - Site 117006, Kyiv
  - Site 117007, Kyiv
  - Site 117012, Kyiv
  - Site 117013, Kyiv
  - Site 117014, Kyiv
  - Site 117016, Kyiv
  - Site 117017, Kyiv
  - Site 117018, Kyiv
  - Site 117020, Kyiv
  - Site 117021, Kyiv
  - Site 117022, Lutsk
  - Site 117003, Ternopil
  - Site 117004, Uzhhorod
  - Site 117010, Uzhhorod
  - Site 117019, Uzhhorod